CLINICAL TRIAL: NCT03206671
Title: B-NHL 2013 - Treatment Protocol of the NHL-BFM and the NOPHO Study Groups for Mature Aggressive B-cell Lymphoma and Leukemia in Children and Adolescents
Brief Title: Treatment Protocol of the NHL-BFM and the NOPHO Study Groups for Mature Aggressive B-cell Lymphoma and Leukemia in Children and Adolescents
Acronym: B-NHL 2013
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Muenster (Other)
Collaborators: Deutsche Krebshilfe e.V., Bonn (Germany) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UKM12_0020; 2013-003253-21 (EudraCT Number)
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Mature B-cell Non-Hodgkin Lymphoma
MeSH Terms: interventions — Cyclophosphamide; Cytarabine; Dexamethasone; Doxorubicin; Vindesine; Etoposide; Ifosfamide; Methotrexate; Prednisolone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- R1/R2 stage I+II (Experimental): Rituximab window + standard chemotherapy without anthracyclines (Vincristine not in R1)
  Interventions: Drug: Rituximab window; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Etoposide; Drug: Ifosfamide; Drug: Methotrexate; Drug: Prednisolone; Drug: Vincristine
- R2 stage III experimental arm (Experimental): Rituximab window + Standard chemotherapy
  Interventions: Drug: Rituximab window; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin hydrochloride; Drug: Etoposide; Drug: Ifosfamide; Drug: Methotrexate; Drug: Prednisolone; Drug: Vincristine
- R2 stage III standard arm (Other): Standard chemotherapy
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin hydrochloride; Drug: Etoposide; Drug: Ifosfamide; Drug: Methotrexate; Drug: Prednisolone; Drug: Vincristine
- R3/R4 rituximab plus arm (Experimental): Rituximab window + standard chemotherapy plus six additional doses of rituximab
  Interventions: Drug: Rituximab window; Drug: Additional doses of Rituximab; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin hydrochloride; Drug: Vindesine Sulfate; Drug: Etoposide; Drug: Ifosfamide; Drug: Methotrexate; Drug: Prednisolone; Drug: Vincristine
- R3/R4 standard arm (Experimental): Rituximab window + standard chemotherapy
  Interventions: Drug: Rituximab window; Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dexamethasone; Drug: Doxorubicin hydrochloride; Drug: Vindesine Sulfate; Drug: Etoposide; Drug: Ifosfamide; Drug: Methotrexate; Drug: Prednisolone; Drug: Vincristine

INTERVENTIONS:
Drug: Rituximab window — Rituximab window (375 mg/m²)
  Arms: R1/R2 stage I+II; R2 stage III experimental arm; R3/R4 rituximab plus arm; R3/R4 standard arm
Drug: Additional doses of Rituximab — 2 doses of Rituximab (375 mg/m²) before the start of the first chemotherapy cycle, 2 doses of Rituximab before the start of the second chemotherapy cycle, 1 dose of rituximab before the start of the third chemotherapy cycle, 1 dose of Rituximab before the start of the forth chemotherapy cycle
  Arms: R3/R4 rituximab plus arm
Drug: Cyclophosphamide — see detailed protocol description
Drug: Cytarabine — see detailed protocol description
Drug: Dexamethasone — see detailed protocol description
Drug: Doxorubicin hydrochloride — see detailed protocol description
  Arms: R2 stage III experimental arm; R2 stage III standard arm; R3/R4 rituximab plus arm; R3/R4 standard arm
Drug: Vindesine Sulfate — see detailed protocol description
  Arms: R3/R4 rituximab plus arm; R3/R4 standard arm
Drug: Etoposide — see detailed protocol description
Drug: Ifosfamide — see detailed protocol description
Drug: Methotrexate — see detailed protocol description
Drug: Prednisolone — see detailed protocol description
Drug: Vincristine — see detailed protocol description

SUMMARY:
The trial B-NHL 2013 is a collaborative prospective, multi-national, multi-center, randomized trial with participating centers of the NHL-BFM group (Austria, Switzerland, Czech Republic, Germany) and the Scandinavian NOPHO group (Denmark, Finland, Norway, Sweden). The aim of the trial is to evaluate the role of rituximab in the treatment of mature aggressive B-cell Non-Hodgkin lymphoma and leukemia (B-NHL and B-AL) in children and adolescents.

The following primary study questions are going to be analyzed:

* the effectiveness (event-free survival) in pediatric patients with very limited mature B-NHL (R1 and R2 stage I and II) of substituting anthracyclines by the rituximab window without compromising survival rates.
* the effectiveness (event-free survival) in pediatric patients with limited mature B-NHL (R2 stage III) randomly assigned to receive the rituximab window plus standard chemotherapy or standard chemotherapy without the rituximab window.
* the effectiveness (event-free survival) and the immune reconstitution (recovery of CD19+ B-cells, IR) in pediatric patients with advanced mature B-NHL/B-AL (R3 and R4 incl. R4 CNS+) treated with BFM-type chemotherapy and randomly assigned schedules of one versus seven doses rituximab.

Secondary study questions will address

* additional parameters for immune reconstitution, lymphocyte subpopulations, immunoglobulin levels, vaccination titers and infection rates
* kinetics of immune reconstitution after treatment
* adverse event and severe adverse event profile
* inter-individual variability of rituximab response
* role of different mechanisms of action of rituximab in advanced B-NHL/B-AL

DETAILED DESCRIPTION:
Risk group stratification:

R1/R2 stage I+II:

* R1: resection status: complete
* R2: resection status: incomplete, stage I and II

R2 III:

- R 2: resection status: incomplete, stage III and LDH < 2 x ULN (according to local reference value for adults)

R3/R4:

* R3: resection status: incomplete, stage III and LDH ≥ 2 x ULN but < 4 x ULN or stage IV/B-AL and LDH < 4 x ULN and CNS negative
* R4: resection status: incomplete, Stage III and LDH ≥ 4 x ULN or stage IV/B-AL and LDH ≥ 4 x ULN and CNS negative
* R4 CNS +: stage IV/B-AL and CNS positive

For patients with very limited disease (R1/R2 stage I/II), the addition of rituximab might allow the omission of anthracyclines without jeopardizing survival rates but reducing acute and long term toxicities. In this treatment arm, it is tested whether the event-free survival is similar to that of the historical control when all patients receive one dose of rituximab as monotherapeutic agent in the rituximab window R five days prior to the start of standard chemotherapy as a substitute for anthracyclines.

For patients with limited disease (R2 stage III) it is tested whether the event-free survival can be improved by adding rituximab to the standard chemotherapy. Two different treatment regimens will be evaluated in a randomized design: Patients in the standard arm will receive the standard chemotherapy. Patients of the rituximab plus arm will receive one dose of rituximab as monotherapeutic agent in the rituximab window R five days prior to the start of standard chemotherapy.

For patients with advanced disease (R3/R4) it is tested whether the event-free survival can be improved by adding rituximab to the standard chemotherapy. Two different rituximab regimens will be evaluated in a randomized design: Patients in the standard arm will receive one dose of rituximab as monotherapeutic agent in the rituximab window R five days prior to the start of standard chemotherapy. Patients of the rituximab plus arm will receive the rituximab window and additional six doses of rituximab added to the first four courses of chemotherapy. In addition the immune reconstitution will be analyzed comparing the effect of the two regimens of rituximab added to standard chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, histological or cytological and immunological proven aggressive mature B-cell Non-Hodgkin lymphoma including Burkitt lymphoma (BL), Burkitt leukemia (B-AL), diffuse large B-cell lymphoma (DLBCL), or mature B-cell NHL not further classified according to current WHO classification124. For rare subtypes (e.g. primary mediastinal large B-NHL, PMLBL, double hit lymphoma or high-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements), consultation of the study center is recommended.
* availability of slides/blocks for reference pathology and international pathology panel (except in cases with immunological and cytomorphological assurance of diagnosis)
* age at diagnosis < 18 years
* diagnostics and treatment in one of the participating centers of the trial
* no previous chemotherapy, no previous lymphoma-directed treatment. No application of steroids for more than two days during the last month
* adequate hepatic, renal and cardiac function, except if alteration is due to lymphoma infiltration. Please contact the study center in case of unclear cases.
* signed informed consent of patient and/or parents/guardians for treatment according to the protocol, participation and transfer of data
* follow-up of at least two years after initial diagnosis is expected
* Certificate of vaccination against hepatitis B or negative serology, defined as

  * evidence of immunization with HBs-antigen negative, anti-HBs positive and anti-HBc negative or
  * negative hepatitis B serology with HBs-antigen negative, anti-HBs and anti- HBc negative

Exclusion Criteria:

* patients with insufficient work up not allowing a correct stratification into the risk groups
* B-cell neoplasia as second malignancy
* any other medical, psychiatric or social condition prohibiting treatment according to the protocol (e.g. previous malignancy, prior organ transplant, HIV infection or AIDS or severe immunodeficiency, etc.)
* participation within a different trial for treatment of B-cell malignancies and/or concurrent treatment within any other clinical trial. Exceptions to this are the NHL-BFM Registry 2012 and trials with different endpoints, involving aspects of supportive treatment which can run parallel to B-NHL 2013 without influencing the outcome of this trial e.g. trials on antiemetics, antibiotics, strategies for psychosocial support etc.
* overt hepatitis B or history of hepatitis B
* hypersensitivity to rituximab or to murine proteins or to any of the other excipients of the Investigational Medicinal Product rituximab (MabThera®) or to ingredients of other IMPs.
* lack of CD20 expression of the lymphoma cells
* pregnancy and lactation

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 650 (Estimated)
Dates: Start 2017-08-03 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) | through study completion, maximal seven years
  EFS is defined as time from start of treatment/randomization up to event or to date of last contact for patients without event. The following occurrences are defined as an event: non-response, progressive disease or relapse, treatment related death, death of any other cause or diagnosis of secondary malignancies.
Immune reconstitution rate (only in R3/R4 patients) | 12 months after start of treatment
  Immune reconstitution rate is defined as percentage of patients achieving age adjusted normal B-cell counts (CD19 positive subpopulations) 12 months after start of treatment.

SECONDARY OUTCOMES:
Overall survival (OS) | through study completion, maximal seven years
  OS is defined as time from start of treatment/randomization up to death of any cause or to date of last contact for patients alive.
Relapse-free survival (RFS) | through study completion, maximal seven years
  RFS is defined as time from start of treatment/randomization up to event or to date of last contact for patients without event. The following occurrences are defined as an event: non-response, progressive disease, or relapse.
Response rate (RR) | after rituximab window on day 5, after prephase (patients with rituximab window on day 10, patients without rituximab window on day 6) and after second course (on an average 5 to 6 weeks after start of treatment)
  Complete response, partial remission, objective effect, stable disease or progressive disease
Adverse event rate | from the first day of protocol defined treatment until two years after start of protocol defined treatment
  Rate of patients with acute toxicity defined as grade III/IV/V AE
Rate of patients achieving normal immunoglobulin level 12 months after start of treatment | 12 months after start of treatment
Time interval to normal immunoglobulin level | through study completion, maximal seven years
Time interval from start of treatment to normal CD19 positive B-cells in the peripheral blood. | through study completion, maximal seven years
Rate of patients with normal lymphocyte subpopulations in the peripheral blood 12 months after start of treatment | 12 months after start of treatment
Interval to normal lymphocyte subpopulations in the peripheral blood. | through study completion, maximal seven years
Rate of infections (defined by CTCAE V4) in the time interval from start of treatment until 24 months after start of treatment | 24 months after start of treatment
Rate of infections (defined by CTCAE V4) in the time interval from start of treatment until immune reconstitution (achievement of age adjusted normal B-cell counts) | through study completion, maximal seven years
Rate of patients with sufficient titers after vaccination one year after start of treatment | 1 year after start of treatment
Immune reconstitution rate (only in R1/R2 patients) | 12 months after start of treatment
  Immune reconstitution rate is defined as percentage of patients achieving age adjusted normal B-cell counts (CD19 positive subpopulations) 12 months after start of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Burkhardt, Prof. Dr. Dr., Principal Investigator — University Hospital Muenster, Klinik für Kinder- und Jugendmedizin - Pädiatrische Hämatologie und Onkologie
Locations (88):
- Austria (6):
  - Univ.Klinik für Kinder- und Jugendheilkunde Graz, Klin. Abteilung für pädiatrische Hämato-Onkologie, Graz
  - Univ.Klinik für Kinder- und Jugendheilkunde Innsbruck, Universitätsklinik für Pädiatrie I, Innsbruck
  - Klinikum Klagenfurt am Wörthersee, Abteilung für Kinder- und Jugendheilkunde, Klagenfurt
  - Kepler Universitätsklinikum, Med Campus IV / Onkologie, Linz
  - LKH Salzburg, Universitätsklinik für Kinder- und Jugendheilkunde, Kinderonkologie, Salzburg
  - St. Anna Kinderspital, Vienna
- Department of Pediatric Hematology and Oncology, University Hospital Motol, Prague, Czechia
- Denmark (4):
  - Børneonkologisk afsnit 303B, Børneafdelingen, Aalborg Universitetshospital Nord, Aalborg
  - Børn og Unge afsnit 4, Børneafdelingen, Aarhus Universitetshospital Skejby, Aarhus
  - Børneonkologisk afsnit 5054, BørneUngeKlinikken, Juliane Marie Centret, Rigshospitalet, Copenhagen
  - Børneonkologisk afsnit H2, H. C. Andersen Børnehospital, Odense Universitetshospital, Odense
- Finland (5):
  - Helsinki University Hospital, Children´s Hospital, Dept of Pediatric Hematology and Oncology, Helsinki
  - Kuopio University Hospital, Paediatric Haematology and Oncology, Kuopio
  - University Hospital of Oulu, Paediatric Haematology and Oncology, Oulu
  - Tampere University Hospital, Paediatric Haematology and Oncology, Tampere
  - Turku University Hospital, Paediatric and Adolescent Haematology and Oncology, Turku
- Germany (53):
  - Universitätsklinikum Aachen, Klinik für Kinder - und Jugendmedizin, Hämatologie / Onkologie, Aachen
  - Klinikum Augsburg, Schwäbisches Kinderkrebszentrum, I. Klinik für Kinder und Jugendliche, Hämatologie / Onkologie, Augsburg
  - Charité Campus Virchow-Klinikum, Zentrum für Kinder- und Jugendmedizin, Abt. Hämatologie / Onkologie, Berg
  - HELIOS Klinikum Berlin-Buch, Kinderklinik, Pädiatrische Hämatologie und Onkologie, Berlin
  - Evangelisches Krankenhaus Bielefeld GmbH, Klinik für Kinder- und Jugendmedizin, Hämatologie und Onkologie, Bielefeld
  - Zentrum für Kinderheilkunde der Universität Bonn, Abt. Päd. Hämatologie / Onkologie, Bonn
  - Städtisches Klinikum Braunschweig gGmbH, Klinik für Kinder- und Jugendmedizin, Station K5 / Päd. Hämato- und Onkologie, Braunschweig
  - Klinikum Bremen-Mitte gGmbH, Prof.-Hess-Kinderklinik,Pädiatrische Onkologie und Hämatologie, Bremen
  - Klinikum der Universität zu Köln, Klinik für Kinder- und Jugendmedizin, Abt. Kinderonkologie und -hämatologie, Cologne
  - Carl-Thieme-Klinikum Cottbus gGmbH, Klinik für Kinder- und Jugendmedizin, Cottbus
  - Vestische Kinderklinik, Universität Witten / Herdecke, Datteln
  - Klinikum Dortmund gGmbH, Klinik für Kinder- und Jugendmedizin, Station K1, Abt. Päd. Onkologie / Hämatologie, Dortmund
  - Universitätsklinik Carl Gustav Carus der TU Dresden, Klinik für Kinder- und Jugendmedizin, Dresden
  - Universitätsklinikum Düsseldorf, Zentrum für Kinder- und Jugendmedizin, Klinik für Päd. Hämatologie und Onkologie, Düsseldorf
  - HELIOS Klinikum Erfurt GmbH, Klinik für Kinder- und Jugendmedizin, Päd. Onkologie / Hämatologie, Erfurt
  - Universitätsklinikum Erlangen, Klinik für Kinder- und Jugendmedizin, Pädiatrische Onkologie / Hämatologie, Erlangen
  - Universitätsklinikum Essen, Zentrum für Kinder- und Jugendmedizin, Hämatologie / Onkologie, Essen
  - Universitätsklinikum Frankfurt, Klinik für Kinder- und Jugendmedizin, Pädiatrische Hämatologie und Onkologie, Frankfurt am Main
  - Universitätsklinikum Freiburg, Zentrum für Kinder- und Jugendmedizin, Klinik IV: Päd. Hämatologie und Onkologie, Freiburg im Breisgau
  - Universitätsklinikum Gießen und Marburg, Standort Gießen, Zentrum für Kinderhämatologie und -onkologie, Giessen
  - Georg-August-Universität Universitäts-Kinderklinik, Pädiatrie I, Göttingen
  - Universitätsklinikum Greifswald KdöR, Klinik und Poliklinik für Kinder- und Jugendmedizin, Abt. Pädiatrische Onkologie und Hämatologie, Greifswald
  - Universitätsklinikum Halle (Saale), Klinik für Kinder- und Jugendmedizin, Pädiatrische Hämatologie / Onkologie, Halle
  - Universitätsklinikum Hamburg Eppendorf, Zentrum für Kinder- und Jugendmedizin, Abt. Pädiatrische Hämatologie und Onkologie, Hamburg
  - Medizinische Hochschule Hannover, Kinderheilkunde, Päd. Hämatologie / Onkologie, Hanover
  - Universitäts-Kinderklinik Heidelberg, Abt. Hämatologie / Onkologie, Heidelberg
  - Gemeinschaftskrankenhaus Herdecke, Kinder- und Jugendmedizin, Päd. Hämatologie / Onkologie, Herdecke
  - Universitätskliniken für Kinder- und Jugendmedizin, Päd. Hämatologie und Onkologie, Geb. 9, Homburg
  - Universitätsklinikum Jena, Klinik für Kinder- und Jugendmedizin, Jena
  - Städtisches Klinikum Karlsruhe gGmbH, Kinderklinik, Station S 24, Karlsruhe
  - Klinikum Kassel Gesundheit Nordhessen Holding AG, Klinik für pädiatrische Hämatologie und Onkologie, Kassel
  - Universitätsklinikum Schleswig Holstein Campus Kiel, Klinik für Allgemeine Pädiatrie, Päd. Onkologie / Hämatologie, Kiel
  - Gemeinschaftsklinikum Mittelrhein Kemperhof, Klinik für Kinder- und Jugendmedizin, Pädiatrische Hämatologie und Onkologie, Koblenz
  - HELIOS Klinikum Krefeld, Zentrum für Kinder- und Jugendmedizin, Päd. Hämatologie/Onkologie, Krefeld
  - Universitätsklinikum Leipzig, Klinik für Kinder und Jugendliche, Abt. Päd. Hämatologie / Onkologie, Leipzig
  - Universitätsklinikum Schleswig Holstein Campus Lübeck, Klinik für Kinder- und Jugendmedizin, Hämatologie und Onkologie, Lübeck
  - Universitätsklinikum Magdeburg A. ö. R., Kinderklinik, Päd. Hämatologie / Onkologie, Magdeburg
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Zentrum für Kinder- und Jugendmedizin, Pädiatrische Hämatologie / Onkologie, Mainz
  - Klinikum Mannheim gGmbH, Universitäts-Kinderklinik, Päd. Onkologie /Hämatologie, Mannheim
  - Johannes Wesling Klinikum Minden, Klinik für Kinder- und Jugendmedizin, Päd. Hämatologie / Onkologie, Station E 22, Minden
  - Klinikum der LMU, Dr. von Haunersches Kinderspital, Pädiatrische Hämatologie / Onkologie, München
  - Klinikum Schwabing, Kinderklinik der TU Päd. Hämatologie / Onkologie, Station 24d, München
  - Universitätsklinikum Münster, Klinik für Kinder- und Jugendmedizin, Abt. Pädiatrische Hämatologie und Onkologie, Münster
  - Diakonie Neuendettelsau, Kliniken Hallerwiese / Cnopf'sche Kinderklinik, Pädiatrische Hämatologie /Onkologie, Nuremberg
  - Klinikum Oldenburg AöR, Zentrum für Kinder- und Jugendmedizin, Abt. Hämatologie / Onkologie, Oldenburg
  - Universitätsklinikum Regensburg, Klinik für Kinder- und Jugendmedizin, Abt. Päd. Hämatologie, Onkologie, SZT, Regensburg
  - Universitätsklinikum Rostock, Kinder- und Jugendklinik, Päd. Hämatologie und Onkologie, Rostock
  - Asklepios Klinik St. Augustin GmbH, Kinder- und Jugendmedizin, Kinder-Hämatologie und Onkologie, Sankt Augustin
  - HELIOS Kliniken Schwerin GmbH, Klinik für Kinder- und Jugendmedizin, Station A1, Schwerin
  - Klinikum Stuttgart, Olgahospital Zentrum für Kinder- und Jugendmedizin Pädiatrie 5 (Onkologie, Hämatologie, Immunologie), Stuttgart
  - Universitätsklinik Tübingen Klinik für Kinderheilkunde und Jugendmedizin, Päd. Hämatologie / Onkologie, Tübingen
  - Universitätsklinikum Ulm, Klinik für Kinder- und Jugendmedizin, Päd. Hämatologie und Onkologie, Ulm
  - Universitätskinderklinik Würzburg, Päd. Onkologie und Hämatologie, Würzburg
- Norway (4):
  - Haukeland University Hospital, National Study Center Norway, Bergen
  - Oslo University Hospital, Rikshospitalet, Oslo
  - University Hospital Northern Norway, Tromsø
  - St Olavs Hospital, Trondheim
- Sweden (6):
  - Sahlgrenska Universitetssjukhuset, Drottning Silvias Barn och Ungdomssjukhus, Barncancercentrum, Gothenburg
  - Universitetssjukhuset i Linköping, Barn och Ungdomsmedicinska kliniken, Barnonkologiska enheten, Linköping
  - Skåne Universitetssjukhus, Barnonkologi, Lund
  - Karolinska Universitetssjukhuset, Astrid Lindgrens Barnsjukhus, Barnonkologen, Stockholm
  - Universitetssjukhus Umeå, Barnonkologiska avdelningen, Barn 3 Norrlands, Umeå
  - Akademiska sjukhuset, Barnavdelningen för blod- och tumörsjukdomar, Uppsala
- Switzerland (9):
  - Kantonsspital Aarau, Kinderklinik, Aarau
  - Universitäts - Kinderspital beider Basel, Basel
  - Ospedale San Giovanni, Reparto die Pediatria, Bellinzona
  - Universitätsklinik für Kinderheilkunde, Pädiatrische Hämatologie/ Onkologie, Inselspital, Bern
  - Hôpital des Enfants, Unité d'Oncologie Hématologie, Geneva
  - Centre hospitalier universitaire vaudois, Unité d'hémato-oncologie pédiatrique, Lausanne
  - Kinderspital Pädiatrische Hämatologie/ Onkologie, Lucerne
  - Ostschweizer Kinderspital, Hämatologie/ Onkologie, Sankt Gallen
  - Universitäts-Kinderspital, Pädiatrische Onkologie, Zurich

IPD SHARING:
Plan to Share IPD: No